CLINICAL TRIAL: NCT00431431
Title: A Multinational, Randomized, Double-Blind, Parallel Group Comparative Trial on the Effects of 2 Years Treatment With Tibolone (1.25 mg Org OD 14) and Raloxifene (60 mg) on Bone Mineral Density in Osteopenic Postmenopausal Women
Brief Title: Comparison of Tibolone and Raloxifene on Bone Mineral Density in Osteopenic Postmenopausal Women (P06090)
Acronym: STEP
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Organon and Co (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Treatment
Other Study IDs: P06090; E-1693
Record Dates: First submitted 2007-02-02; First posted 2007-02-05 (Estimated); Last update posted 2024-08-15 (Actual); Status verified 2022-02

CONDITIONS: Osteopenia
MeSH Terms: conditions — Bone Diseases, Metabolic | interventions — tibolone

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- 1 (Experimental): tibolone
  Interventions: Drug: tibolone
- 2 (Active Comparator): raloxifene
  Interventions: Drug: raloxifen

INTERVENTIONS:
Drug: tibolone — 2 years treatment with tibolone (1.25 mg Org OD-14)
  Arms: 1
Drug: raloxifen — 2 years treatment with raloxifene (60 mg)
  Arms: 2

SUMMARY:
Both tibolone and raloxifene have been demonstrated to prevent postmenopausal bone loss. During treatment with tibolone bone mineral density (BMD) of the spine has been shown to be increased between 1.8 and 5.8 % above baseline in two years, depending on the population studied. Since treatments aimed at prevention should ideally be used long-term, compliance with the treatment is crucial. Efficacy of and compliance with the two treatments will be measured and evaluated.

ELIGIBILITY:
Inclusion Criteria:

* Only subjects who give voluntary written informed consent, and who are willing and able to make reasonable efforts to observe all clinical trial requirements are to be enrolled.
* Subjects will be osteopenic but otherwise healthy postmenopausal women, from 60 to 79 years of age (inclusive) at entry.
* Screening BMD of the lumbar vertebrae (L1-L4) must be between -2.5 SD and

  * 1.0 SD of the T-score.
* Subjects should have a Body Mass Index (BMI) >19 and < 30 kg/m2.

Exclusion Criteria:

* Spinal X -ray with symptomatic vertebral fracture (more than 20% reduction in expected vertebral height).
* History of bilateral hip replacements.
* Subjects who are not ambulatory.
* History or presence of any malignancy, except non-melanoma skin cancers.
* TVUS double wall thickness > 4 mm, or any other undiagnosed abnormalities visualized by TVUS.
* Abnormal cervical Pap smear result
* Undiagnosed abnormal (in the investigator's opinion) vaginal bleeding in the past year prior to screening.
* Mammography or physical examination finding that is suspicious of malignancy.
* Uncontrolled hypertension
* Bone disease other than osteoporosis such as Paget's disease, osteomalacia or bone metastases.
* Drinking more than 4 glasses of alcohol containing drinks per day.
* Smoking more than 20 cigarettes a day.
* Current or recent prolonged use of hepatic microsomal enzyme-inducing anticonvulsant medication or other drugs known to interfere with or otherwise alter the pharmacokinetics of steroids.
* Treatment with anabolic steroids, calcitonin or raloxifene within the last 6 months.
* Treatment with alendronate and risedronate more than 6 months. If treatment duration was less than 6 months a wash-out period of 12 months is necessary.
* Treatment with etidronate for 1 year a wash-out period of 6 months is necessary. If treatment period of more than 1 year a wash -out period of 12 months is necessary.
* Treatment with oral estrogen and/or progestin therapy (including contraceptives) or transdermal therapy and local estrogen applications within 6 months prior to screening/baseline BMD measurements (i.e. the wash -out period of 6 months must have been completed before the screening / baseline BMD assessments are made). A 20-week wash-out for injections of MPA-containing contraceptives (e.g. Depo-Provera®) is required.
* Ever use of estrogen and/or progestin containing implants.
* The use of cholesterol-lowering medicine cholestyramine or colestipol.
* Subjects with a change in thyroid medication within the last 6 weeks prior to screening.
* Subjects who have had fluoride treatment for 2 weeks or more (> 2 mg/day fluorideion) at any time (NaF tablets for caries prevention is allowed).
* Subjects who have undergone systemic glucocorticoid treatment (> 5 mg prednisone or equivalent/day) for more than one month within the past 6 months (prior to BMD screening assessments).
* Subjects who are receiving or require medication for the treatment of osteoporosis except Calcium / Vit D.
* The use of coumarin products.
* Type I diabetes mellitus.
* Presence or history of thromboembolic disorders.
* Serious decompensated renal or liver disease.
* Abnormal laboratory values
* Any condition or disease that could result in altered absorption, excessive accumulation, impaired metabolism, or altered excretion of the investigational product.

Ages: 60 Years to 79 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 324 (Actual)
Dates: Start 2000-07-31 (Actual); Primary Completion 2005-02-15 (Actual); Study Completion 2005-02-15 (Actual)

PRIMARY OUTCOMES:
Measure BMD to evaluate the effects of treatment on bone mineral density of the lumbar vertebrae L1-L4 | At screening, after 52 weeks and 104 weeks

SECONDARY OUTCOMES:
To measure the effects on hot flushes by using diary booklets | Throughout trial and up to week 52
To measure the economic impact during the whole trial period by using Medical resource utilization forms | Baseline and week 52 and 104
Bone mineral density of the total hip | At screening, week 52 and week 104
A vaginal smear to determine vaginal atrophy | At screening, week 52 and week 104
Biochemical markers of bone metabolism | At baseline, week 12, week 24, week 52 and week 104
McCoy Female Sexuality Questionnaire, Short -Form to assess sexual functioning, Women's Health Questionnaire to assess quality of life, Health Utility Index Mark 2 and 3 (HUI2/HUI3) to confirm the health status | At baseline, week 12, week 24, week 52 and week 104

REFERENCES:
- [Result] Delmas PD, Davis SR, Hensen J, Adami S, van Os S, Nijland EA. Effects of tibolone and raloxifene on bone mineral density in osteopenic postmenopausal women. Osteoporos Int. 2008 Aug;19(8):1153-60. doi: 10.1007/s00198-007-0545-3. Epub 2008 Feb 7. PMID 18256777